CLINICAL TRIAL: NCT05973942
Title: Population Impact of Wingman-Connect Implemented by the US Air Force
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Peter A. Wyman, Professor, University of Rochester
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00008550
Record Dates: First submitted 2023-07-25; First posted 2023-08-03 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Suicide Prevention
Keywords: military; suicide rates
MeSH Terms: conditions — Suicide Prevention

STUDY DESIGN:
Intervention Model Description: Stepped Wedge. The US Air Force is implementing Wingman-Connect (Wyman et al, 2020) in collaboration with University of Rochester researchers in the context of First Term Airmen Classes (FTAC) across 8 operational bases. The AF has agreed to stagger implementation based on randomization informed by a stepped-wedge design. Wingman-Connect training will be rolled out at 8 USAF bases in pairs at 3 month intervals and will continue for a total of 51 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wingman-Connect (Experimental): Wingman-Connect (Wyman et al., 2020) uses a network health theoretical framework to strengthen two suicide-protective functions of social networks: 1) Strengthening positive social bonds, and 2) Building healthy norms that incentivize adaptive coping. Training will be delivered in First Term Airmen classes among all Airmen arriving at base during the study period.
  Interventions: Behavioral: Wingman-Connect

INTERVENTIONS:
Behavioral: Wingman-Connect — Training occurs in three 2-hr blocks over several days. Targeted Skills focus on protective factors (Four Cores) supportive of mental health, theoretically linked to reduced suicide risk, and essential to an Airmen's job success: (1) Healthy relationships and accountability spanning USAF and family/intimate relationships (Kinship); (2) Meaning and value in work and life (Purpose), (3) Informal and formal help-seeking (Guidance); and (4) Activities that give strength and balance emotions (Balance). Activities progress from individual to group skill-building activities. Kinship modules at operational base (FTAC) expand focus on growing and sustaining relationships with intimate partners, friends, and family; and Guidance more on senior mentors at work.

SUMMARY:
This study involves collection of implementation data and analysis of USAF de-identified administrative data on base-level suicide attempt rates following US Air Force (USAF) delivery of Wingman-Connect training at 8 operational AF bases, as part of a force-wide scale out of the program. Implementation of Wingman-Connect by the USAF will occur over 51 months. The AF has agreed to stagger implementation based on a randomized stepped-wedge design. Once Wingman-Connect has been initiated at each base, all entering first-term Airmen will receive Wingman-Connect, with ~17,400 total Airmen receiving Wingman-Connect across all bases.

Implementation. The study will directly collect data from USAF prevention personnel who are involved in the delivery of the intervention to measure fidelity and measure implementation barriers and facilitators. These base-level data are essential to test Wingman-Connect impact on suicide attempt rates in a general USAF population, to study Wingman-Connect diffusion, and to refine implementation processes and tools.

Suicide Rates. Bases routinely provide their base-wide suicide attempt rates to the Air Force Medical Readiness Agency (AFMRA). AFMRA will provide these routinely-collected aggregate administrative data to this study in order to analyze changes in base-level suicide attempt rates (USAF administrative data) among the 8 bases.

DETAILED DESCRIPTION:
The US Air Force is putting into regular practice the Wingman-Connect Program in the context of First Term Airmen Courses (FTAC) across all 68 operational bases, beginning with 8 bases in two Major Commands (AFGSC, AMC). University of Rochester researchers will provide facilitator training and ongoing fidelity monitoring. Wingman-Connect uses a network health theoretical framework to strengthen two suicide-protective functions of social networks: 1) Strengthening positive social bonds, and 2) Building healthy norms that incentivize adaptive coping. Implementation of Wingman-Connect by the USAF will occur over 51 months. The AF has agreed to stagger implementation based on a randomized stepped-wedge design. Pairs of bases will begin implementation of the program in all FTAC at 3 months intervals and continue over a 51 month total period. Data collection will begin with the start of implementation at each base.

Implementation. The study will directly collect data from USAF prevention personnel who are involved in the delivery of the intervention to measure fidelity and measure implementation barriers and facilitators at each location. Prevention personnel will complete measures every 6 months. Due to turnover of personnel (training site administrators every 6 months) we anticipate 8-12 individual respondents per site across the study period, and 4-6 respondents at each site per data point, for a possible total of N=96 respondents. These participants are also expected to reflect the demographics of the USAF as a whole. Measures will include base climate, uptake of program, USAF implementers' fidelity delivering Wingman-Connect and engagement in training/technical support.

Suicide Rates. Bases routinely provide their base-wide suicide attempt rates to the Air Force Medical Readiness Agency (AFMRA). To test effectiveness of Wingman-Connect delivered by the USAF on these bases, the AFMRA will provide these routinely-collected aggregate administrative data to this study in order to analyze changes in base-level suicide attempt rates (USAF administrative data) among the 8 bases. AFMRA will provide suicide attempt and suicidal behavior data for Airmen of E1-E4 ranks (incoming first term Airmen) on each base every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Data from bases in the Air Force Global Strike Command (AFGSC) & Air Mobility Command (AMC) MajComs.
* 96 implementers (4-5 per base over at each data point, and 8-12 respondents per site across the study period)

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17400 (Estimated)
Dates: Start 2024-08-13 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Total Number Base level suicide attempts among Ranks E1-4 | 4 years
  Suicide attempt data for the total population of junior Airmen on each base will be collected from the Air Force Medical Readiness Agency (AFMRA) through our study sponsor Office of Integrated Resilience (HAF/A1Z). Suicide attempt data is compiled using ICD-10 codes for patient encounters across multiple sources including records from direct-care within Air Force medical systems (CAPER, SIDR, M2).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data on base-level suicide attempts will be made available at the NIMH Data Archive (NDA). Any coding used to manipulate data (create categories, scales) will be done in either SPSS or R and this code will also be provided via NDA or github.
Supporting Information: Study Protocol, SAP
Time Frame: All data will be deposited to NDA starting 12 months after the award begins and will be deposited every six months thereafter following the usual NDA data submission dates.
Access Criteria: To request access of the data, researchers will use the standard processes at NDA, and the NDA Data Access Committee will decide which requests to grant. The standard NDA data access process allows access for one year and is renewable.
URL: https://nda.nih.gov/

REFERENCES:
- [Background] Wyman PA, Pickering TA, Pisani AR, Cero I, Yates B, Schmeelk-Cone K, Hendricks Brown C, Gibbons RD, Simonson J, Pflanz SE. Wingman-Connect Program increases social integration for Air Force personnel at elevated suicide risk: Social network analysis of a cluster RCT. Soc Sci Med. 2022 Mar;296:114737. doi: 10.1016/j.socscimed.2022.114737. Epub 2022 Jan 22. PMID 35131614
- [Background] Wyman PA, Pisani AR, Brown CH, Yates B, Morgan-DeVelder L, Schmeelk-Cone K, Gibbons RD, Caine ED, Petrova M, Neal-Walden T, Linkh DJ, Matteson A, Simonson J, Pflanz SE. Effect of the Wingman-Connect Upstream Suicide Prevention Program for Air Force Personnel in Training: A Cluster Randomized Clinical Trial. JAMA Netw Open. 2020 Oct 1;3(10):e2022532. doi: 10.1001/jamanetworkopen.2020.22532. PMID 33084901